CLINICAL TRIAL: NCT03933995
Title: Follow up Study(Phase 1) to Evaluate Safety of Autologous Bone Marrow Derived Mesenchymal Stem Cell in Erectile Dysfunction
Brief Title: Follow up Study(Phase 1) to Evaluate Safety of Autologous Bone Marrow Derived MSCs in Erectile Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMC-P-09
Record Dates: First submitted 2019-04-15; First posted 2019-05-01 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mesenchymal stem cell: Long-term follow up of Mesenchymal stem cell group
  Interventions: Other: no Intervention

INTERVENTIONS:
Other: no Intervention — no Intervention

SUMMARY:
This is a 5year (+-30 days) long term follow up study to evaluate the safety of autologous bone marrow derived mesenchymal stem cell in erectile dysfunction subject who participated in and completed the Phase 1 trials (refer to ClinicalTrials.gov.Identifier: NCT02344849).

DETAILED DESCRIPTION:
This is a 5year (+-30 days) long term follow up study to evaluate the safety of autologous bone marrow derived mesenchymal stem cell in erectile dysfunction subject who participated in and completed the Phase 1 trials (refer to ClinicalTrials.gov.Identifier: NCT02344849).

This trial is planned to evaluate the safety of autologous bone marrow derived mesenchymal stem cell in patients with erectile dysfunction subject. Subjects who signed this follow-up observation informed consent form will participate in a safety assessment (tumor marker test, Serious Adverse Events, cancer incidence, recurrence of prostate cancer and vital sign).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who treated with Mesenchymal stem cell and enrolled the phase 1 study(NCT02344849).
2. Subjects who can agree to participate in the long term observation study by oneself.

Exclusion Criteria:

* Not Applicable

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who treated with Mesenchymal stem cell and enrolled the phase 1 study(NCT02344849).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation assessed by Tumor Marker Test. | 5 year(+-30 days)
  Tumor Marker Test(reported in ng/mL): PSA, AFP, CEA Tumor Marker Test is optional item, not mandatory.
  In this study, tumor markers divided into which are classified as "Normal / Not clinical significant / Clinical significant" abnormalities and analysis the frequency and proportion.
Safety Evaluation assessed by Serious Adverse Events, cancer incidence and recurrence of prostate cancer. | 5 year(+-30 days)
  Safety Evaluation assessed by Tumor Marker Test, patient reporting and vital signs
  For each subject who has had one or more serious adverse events since the ongoing clinical trial, the severity of the adverse reaction should be provided for each causal relationship, and the incidence of serious adverse events should be analyzed.
Safety Evaluation assessed by Vital Signs. | 5 year(+-30 days)
  Vital Sign : Blood pressure(reported in mmHg), Pulse(reported in time/min) Vital Sign is optional item, not mandatory.
  The vital sign values obtained from this study were compared for each group. Baseline statistics (mean, standard deviation, median, maximum, and minimum) are presented, and clinically significant figures are summarized and presented based on the normal range for each value.

CONTACTS AND LOCATIONS:
Overall Officials: Chungsu Kim, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided